CLINICAL TRIAL: NCT03037957
Title: A Multi-Site Clinical Evaluation of the ARIES Group A Strep Assay in Symptomatic Patients
Status: Completed | Type: Observational
Sponsor: Luminex Corporation (Industry)
Responsible Party: Sponsor
Organization: Luminex Molecular Diagnostics (Industry)
Other Study IDs: LMA-GAS-01-CS-006
Record Dates: First submitted 2017-01-03; First posted 2017-01-31 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Pharyngitis Bacterial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A Strep Assay
  Interventions: Device: ARIES Group A Strep Assay

INTERVENTIONS:
Device: ARIES Group A Strep Assay

SUMMARY:
A multi-center evaluation to assess the diagnostic sensitivity and specificity of the ARIES Group A Strep Assay will be established through a method comparison using prospectively collected, de-identified, clinical samples collected during the enrollment period.

ELIGIBILITY:
Inclusion Criteria:

* Patient and/or patient's legal guardian is willing and able to give informed consent and/or assent for extra research sample.
* The subject's specimen is a throat swab in Liquid Amies based transport medium.
* The specimen is from an adult or pediatric, male or female subject who is either hospitalized, admitted to a hospital emergency department, visiting an outpatient clinical or resident of a long term care facility.
* The specimen is from a patient for whom a requisition has been made for Group A Strep testing
* The specimen is from a patient exhibiting clinical signs and symptoms of pharyngitis consistent with Group A Strep infection.
* The specimen was received in good condition (no leakage or drying of the specimen).
* The specimen volume is ≥ 850 µL.

Exclusion Criteria:

* The specimen is from a patient who did not provide informed consent/assent.
* The specimen is not a throat swab collected in Liquid Amies based transport medium.
* The specimen is from a patient who is undergoing antibiotic treatment.
* The specimen was not properly collected, transported, processed or stored according to the instructions provided by the Sponsor in Section 9 below.
* The specimen volume is < 850 µL.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting with signs and symptoms of pharyngitis for which their doctors ordered a Group A Strep test.
Sampling Method: Non-Probability Sample
Enrollment: 704 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Clinical performance (sensitivity/specificity) for Group A Strep Assay | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Dunn, Study Director — Luminex Corporation
Locations (5):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Sacred Heart Hospital, Pensacola, Florida
  - Children's Mercy Hospital, Kansas City, Missouri
  - Advanced Pediatrics Research, Vienna, Virginia
  - Marshfield Labs, Marshfield, Wisconsin